CLINICAL TRIAL: NCT04453111
Title: Efficacy of Bone-marrow-derived and Placenta-derived Multipotent Mesenchymal Stem / Stromal Cells for Osteoarthritis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Cell Therapy (Industry)
Collaborators: The Institute of Traumatology and Orthopedics of NAMS of Ukraine (Unknown); Kyiv City Clinical Hospital № 6 (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #7/09.26.2018
Record Dates: First submitted 2020-06-15; First posted 2020-07-01 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Knee Osteoarthritis
Keywords: BM-MMSCs;; P-MMSCs;; Hyaluronic Acid
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: Experimental: HA + stem cells therapy Experimental Group 1: three intra-articular injection of allogeneic P-MMSCs with up to 2•107cells (target dose up to 6•107 cells) with 20 mg Hyaluronic Acid at 4-weeks intervals - 15 patients Experimental Group 2: three intra-articular injection of autologous BM-MMSCs up to 2•107cells (target dose up to 6•107 cells) with 20 mg Hyaluronic Acid at 4-weeks intervals - 15 patients Control Group: three intra-articular injection of 20 mg Hyaluronic Acid, no cell therapy - 15 patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hyaluronic Acid (HA) + P-MMSCs (Experimental): Experimental Group 1: Three intra-articular injection of allogeneic P-MMSCs up to 2•107cells (target dose up to 6•107 cells) with 20 mg Hyaluronic Acid at 4-weeks intervals - 15 patients
  Interventions: Biological: Placenta-derived MMSCs; Drug: Hyalgan 20 mg in 2 ML Prefilled Syringe
- Hyaluronic Acid (HA) + BM-MMSCs (Experimental): Experimental Group 2: Three intra-articular injection of autologous BM-MMSCs up to 2•107cells (target dose up to 6•107 cells) with 20 mg Hyaluronic Acid at 4-weeks intervals - 15 patients
  Interventions: Biological: Bone marrow-derived MMSCs; Drug: Hyalgan 20 mg in 2 ML Prefilled Syringe
- Hyaluronic Acid (HA) (Active Comparator): Three intra-articular injection of 20 mg Hyaluronic Acid - 15 patients
  Interventions: Drug: Hyalgan 20 mg in 2 ML Prefilled Syringe

INTERVENTIONS:
Biological: Placenta-derived MMSCs — Cryopreserved placenta-derived multipotent mesenchymal stem / stromal cells
  Other Names: P-MMSCs
  Arms: Hyaluronic Acid (HA) + P-MMSCs
Biological: Bone marrow-derived MMSCs — Cryopreserved bone marrow-derived multipotent mesenchymal stem / stromal cells
  Other Names: BM-MMSCs
  Arms: Hyaluronic Acid (HA) + BM-MMSCs
Drug: Hyalgan 20 mg in 2 ML Prefilled Syringe — Hyaluronic Acid 20 mg
  Other Names: HA

SUMMARY:
To define the clinical effects of intra-articular transplantation of bone-marrow-derived (BM-MMSCs) and placenta-derived multipotent mesenchymal stem / stromal cells (P-MMSCs) for knee osteoarthritis.

DETAILED DESCRIPTION:
Multipotent mesenchymal stem / stromal cells (MMSCs) of different origin are the novel therapeutic agents that can slow down cartilage degeneration, improve reparation and ultimately prevent joint prosthetics. MSCs are capable to direct differentiation into chondrocytes, produce cytokines and growth factors with immunomodulatory and anti-inflammatory effects, stimulate angiogenesis, as well as induce chemotaxis of endogenous progenitors. Bone marrow-derived and placenta-derived MMSCs can be considered the most promising source for cell therapy of joints disorders according to availability, safety and expected therapeutic efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of knee osteoarthritis.
2. Age: 18 to 75 years old.
3. Kellgren-Lawrence Grade 2 or 3 according to X-ray imaging.
4. Knee pain.
5. Written informed consent

Exclusion Criteria:

1. Age <18 or >75 years of age by time of infusion.
2. Participation in an on-going investigational therapeutic or device trial 30 days of consent.
3. Rheumatoid arthritis.
4. Psoriatic arthritis.
5. Juvenile idiopathic arthritis.
6. Gout.
7. Infectious arthritis.
8. Osteomyelitis.
9. Osteonecrosis.
10. Inflammatory arthritis.
11. Chondropathy.
12. Joint contracture.
13. Arthroplasty.
14. Arthroscopy within 6 months prior to study entry.
15. Intra-articular injection within 3 months prior to study entry.
16. Hormone intake.
17. Antiaggregants and anticoagulants intake.
18. Immunosuppressants intake.
19. Allergy to hyaluronic acid.
20. History of organ or cell transplantation.
21. Hematologic abnormality evidenced by hematocrit < 25%, white blood cell < 2,500/ul or platelet count < 100,000/ul.
22. Active infection.
23. Positive for HIV antigen.
24. History of hepatitis B, hepatitis C.
25. History of malignancy in the last 5 years prior to study entry.
26. Active tumors.
27. History of myocardial infarction.
28. History of stroke.
29. Renal failure with chronic hemodialysis.
30. Liver Cirrhosis (ICGR 15 >30%).
31. Chromosomal abnormality.
32. Peripheral nervous system disorders.
33. Cognitive or language barriers that prohibit obtaining informed consent or any study elements.
34. History of drug abuse or alcohol abuse, or documented medical, occupational, or legal problems arising from the use of alcohol or drugs within the past 24 months.
35. Pregnant/nursing women or women of child-bearing potential.
36. Other condition that limits lifespan to < 1 year.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events and changes in physical examinations, vital signs and the results of clinical lab tests. | 12 months
  Treatment-related adverse events

SECONDARY OUTCOMES:
Physical function improvement measured by Western Ontario and McMaster Universities Arthritis Index (WOMAC). | 12 months.
  Change in joint function from baseline WOMAC assessment. The WOMAC used a scoring scale of 0-4 (lower scores indicate lower levels of symptoms or physical disability). The higher the score, the higher the amount of pain, stiffness, and a high level of functional limitations.
Radiographic evidence. Whole-Organ Magnetic Resonance Imaging Score (WORMS) | 12 months
  Change in cartilage thickness of the knee using MRI
Quality of Life (QOL) assessment | 12 months
  Change in scores on the QOL
The Visual Analog Scale (VAS) assessment | 12 months
  VAS - measure of pain intensity. The scale is most commonly anchored by "no pain " (score of 0) and "worst imaginable pain" (score of 10).

CONTACTS AND LOCATIONS:
Overall Officials: Peter Nemtinov, MD, Study Director — Institute of Cell Therapy
Locations (1):
- Institute of Cell Therapy, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holiuk Y, Birsa R, Bukreieva T, Nemtinov P, Kyryk V, Ustymenko A, Mazevych V, Sokolov M, Lobyntseva G, Shablii V. Effectiveness and safety of multiple injections of human placenta-derived MSCs for knee osteoarthritis: a nonrandomized phase I trial. BMC Musculoskelet Disord. 2025 Apr 26;26(1):418. doi: 10.1186/s12891-025-08664-2. PMID 40281581